CLINICAL TRIAL: NCT04379115
Title: Optimization of Non-Invasive Brain Stimulation for Treatment of Addiction
Brief Title: Optimization of NIBS for Treatment of Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20190760
Record Dates: First submitted 2020-04-21; First posted 2020-05-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Opioid-use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: single-center, double-blinded, placebo controlled, randomized study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (tDCS) + Active TUS (Active Comparator): Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS)
  Interventions: Device: Active Comparator: Active tDCS + Active TUS
- Sham (tDCS) + Sham TUS (Sham Comparator): Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  Interventions: Device: Sham Comparator: Sham tDCS + Sham TUS

INTERVENTIONS:
Device: Active Comparator: Active tDCS + Active TUS — Device: Active comparator device: Active transcranial Direct Current Stimulation (tDCS). Subjects will receive 20 minutes of active tDCS. During each Active stimulation session, stimulation will be applied for the full 20 minutes.
  Device: Active comparator device: Active Transcranial Ultrasound (TUS). Subjects will receive 20 minutes of active Transcranial Ultrasound (TUS). During active stimulation the (TUS) will be active for the full 20 minutes.
  Arms: Active (tDCS) + Active TUS
Device: Sham Comparator: Sham tDCS + Sham TUS — Device: SHAM Comparator Device: transcranial Direct Current Stimulation (tDCS) Subjects will receive 20 minutes of sham tDCS. In the sham group, the tDCS device will not be active for the full 20 minutes.
  Device: Transcranial Ultrasound (TUS) Subjects will receive 20 minutes of sham TUS. During sham stimulation the ultrasound will not be active for the full 20 minutes.
  Arms: Sham (tDCS) + Sham TUS

SUMMARY:
The purpose of this study is to assess the effects of transcranial Direct Current Stimulation (tDCS) applied in conjunction with Transcranial Ultrasound (TUS) for the treatment of addiction in opiate use disorder with chronic pain. The investigators hypothesize that there will be a decrease in drug use and improved psychosocial assessments with active stimulation, when compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent to participate in the study.
2. 18 to 85 years old.
3. Having a diagnosis of OUD, in the setting of CP:

   * OUD of more than 6 months duration as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-5) [64] and a positive urine toxicology screen.
   * or OUD patients who still feel craving or have not received more than 60 mg of methadone/day from the Methadone program.
4. Lives in the immediate area with no plans to relocate

Exclusion Criteria:

1. The subject is pregnant.
2. Recently started on antiepileptic drug therapy.
3. History of illegal stimulant use as demonstrated by urine toxicology.
4. . Ingestion of poppy seeds or herbal teas containing Papaveris Fructus (may cause a positive opiate test for morphine, codeine [66, 67]).
5. History of neurological disorders involving stroke, brain tumors, or epilepsy as self- reported (note patients will also be evaluated via electroencephalography (EEG) at baseline 1 week prior to stimulation and any patient showing abnormal EEG activity will be removed)).
6. History of unexplained fainting spells as self-reported.
7. History of head injury resulting in more than a momentary loss of consciousness as self-reported.
8. History of brain surgery as self-reported.
9. Contraindications to tDCS applied in conjunction with TUS:

   * Metal in the head, or
   * Implanted brain medical devices.
10. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory (BDI), PHQ-9≥10).
11. Active malignancy.
12. History of suicidal behavior or suicide attempts.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-04-04 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in drug use from baseline. | Measured for approximately 6 weeks
  American Pain Foundation Pain/Medication Diary is used to monitor Drug Use overtime after stimulation for approximately 6 weeks.

SECONDARY OUTCOMES:
Changes in the Verbal Rating Scale (VRS) for Pain | Measured for approximately 6 weeks
  Changes in VRS for Pain will be measured in order to determine if tDCS + ESSTIM is effective in reducing the pain of subjects with Chronic Pain (CP) and Opioid Use Disorder(OUD) when compared to the SHAM group.Verbal Rating Scale (VRS) for Pain is a categorical scale of pain with categories: none, mild, moderate, severe pain intensity.
Changes in pain as measured by the Visual Analog Scale (VAS) | Measured for approximately 6 weeks
  Changes in VAS for Pain will be measured in order to determine if tDCS + ESSTIM is effective in reducing the pain of subjects with Chronic Pain (CP) and Opioid Use Disorder(OUD) when compared to the SHAM group.Visual Analog Scale (VAS) for Pain will assess a patient's pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable).
Safety measures | Measured for approximately 6 weeks
  The investigators will measure safety through a standardized neurological exam, which will include the assessment of cognitive domains including memory, attention, mood (scaled as normal or abnormal).
Study 36-Item Short Form (SF-36) | Measured for approximately 6 weeks
  This is a health survey using a scale from 0 (worst) to 100 (best)
Patient Health Questionnaire (PHQ-9) | Measured for approximately 6 weeks
  This questionnaire screens for depression with a score of 0 (best) to 27 (worst)
Electroencephalography (EEG) recording: | Measured for approximately 6 weeks
  previous: EEG recording: On the first baseline visit, on the first day of Week 1, at the end of each stimulation week, and at the follow up visits. EEG recordings will be taken to monitor changes in power in different frequency bands including (theta, alpha, beta and gamma) for 20 min.
Ultimatum Game: | Measured for approximately 6 weeks
  This task evaluates reward, salience and executive network behavioral correlates
Risk Task: | Measured for approximately 6 weeks
  The task is designed to analyze the relationship between prediction and reward (and penalty) is associated with the choice of the least likely outcome, and the smallest reward (and penalty).
Inhibitory Control Task: | Measured for approximately 6 weeks
  We will assess the interaction between reward processing (via the presence or absence of reward) and mechanisms of inhibitory control.
Opioid Cue-Exposure Task for Craving Assessment: | Measured for approximately 6 weeks
  A set of randomized videos showing scenes of people using opioids will aid assessment of craving.
Hair follicle drug test | Measured for approximately 6 weeks
  A hair follicle drug test screens for illicit drug use and the misuse of prescription medication. The sample is then analyzed for signs of drug use over 90 days. The results will be measured as positive or negative.
National Institute on Drug Abuse (NIDA)-Modified ASSIST (NM ASSIST) | Measured for approximately 6 weeks
  Clinician's Screening Tool for Drug Use in General Medical Settings which implements a scale from 0-3 "Low Risk", 3-26 " Moderate Risk", and 27+ "High Risk"
Obsessive-Compulsive Drinking/Drug Use Scale (OCDS) | Measured for approximately 6 weeks
  This measure reflects obsessionality and compulsivity related to craving and drinking behavior with a total score ranging from 0 to 64 (with 64 being the worst).
15-item Barrett Impulsivity scale | Measured for approximately 6 weeks
  15-item Barrett Impulsivity scale is used to measure impulsivity with a total score ranging from 15 to 60 (with 15 lower level of impulsivity and 60 higher levels of impulsivity.
National Institute on Drug Abuse (NIDA) Quick Screen | Measured for approximately 6 weeks
  The NIDA Quick Screen is a validated instrument designed to assist providers in screening adults for substance use which has a yes/no scale (with "no" being best and "yes" being worse)
Urine drug test | Measured for approximately 6 weeks
  A Urine drug test screens for illicit drug use and the misuse of prescription medication. The sample is then analyzed for signs of drug use during the past few days. The results will be measured as positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ciro R Estebanez, MD PhD, Principal Investigator — University Hospitals Cleveland Medical Center/ Case Western Reserve University
Locations (3):
- United States (3):
  - University of Illinois Health/ University of Illinois at Chicago, Hinsdale, Illinois
  - Spaulding Rehabilitation Hospital - 5th Floor - Neuromodulation Center, Cambridge, Massachusetts
  - University Hospitals Cleveland Medical Center/ Dahms Clinical Research Unit, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No